CLINICAL TRIAL: NCT01880034
Title: Availability of Lipid Emulsion to Regional Anesthesia Programs at US Academic Anesthesia Departments
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-0324
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Local Anesthetic Systemic Toxicity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Regional Anesthesia Section Heads: This group will consist of Regional Anesthesia Section Heads at anesthesia residency training programs.
  Interventions: Other: Lipid Emulsion Survey

INTERVENTIONS:
Other: Lipid Emulsion Survey

SUMMARY:
Significant data exists to suggest that lipid emulsion administration in the setting of local anesthetic toxicity has the potential to be life-saving. Unfortunately, a variety of potential barriers exist to routine lipid emulsion administration for those performing regional anesthesia including drug availability, drug cost and drug location. Inadequate training or lack of established protocols also have the potential to negatively impact patient outcomes. A previous study by Toledo et al (Availability of lipid emulsion in United States obstetric units. Anesth Analg 2013;116:406-408.) evaluated lipid emulsion availability on obstetric units and found that it was nearly universally available.

The Accreditation Council for Graduate Medical Education (ACGME) publishes a list of contact information for each anesthesia institution that engages in resident training. Investigators will contact these institutions by phone or email to obtain contact information for their regional anesthesia program director. In the absence of a program director, investigators will send a survey and consent information via email to the faculty physician most involved in regional anesthesia. Survey completion instructions (survey itself to be completed on Qualtrics Survey Hosting Service) and copy of the study consent form will be attached to the initial contact email. The study consent form will contain a description of the study itself. Survey participants will be allowed time to complete their survey in private at their discretion. Non-responders will receive two follow-up emails at one month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Regional Anesthesia Section heads at academic anesthesia institutions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Regional Anesthesia Section heads at academic anesthesia institutions.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Is lipid emulsion available at all locations where regional anesthesia is practiced in your institution? | Two months
  Survey options include
  1. Yes, lipid emulsion is available in the room where regional anesthesia is performed.
  2. Yes, lipid emulsion is available in a near-by pharmacy
  3. Yes, lipid emulsion is available in a central pharmacy
  4. No, lipid emulsion is not available in all locations where regional anesthesia is performed

SECONDARY OUTCOMES:
If lipid emulsion is available to those practicing regional anesthesia at your institution, how long would it take to obtain it? | Two Months.
  Possible responses include:
  * Lipid emulsion is not available at our institution.
  * Less than 10 minutes
  * 10-30 minutes
  * More than 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States